CLINICAL TRIAL: NCT04874389
Title: Multimodal Screening and Diagnostic Approaches to Brain Trauma in Performance Populations
Brief Title: Multidimensional Classification of Mild Traumatic Brain Injury (mTBI)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Clea Tucker (Other)
Responsible Party: Sponsor-Investigator, Clea Tucker, Assistant Professor; Doctor of Physical Therapy, California State University, Los Angeles
Organization: California State University, Los Angeles (Other)
Other Study IDs: 1502994
Record Dates: First submitted 2021-04-30; First posted 2021-05-05 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Mild Traumatic Brain Injury
Keywords: brain oxygenation; functional multimodal assessment; dual tasking; traumatic brain injury; balance; gait; cognition
MeSH Terms: conditions — Brain Concussion; Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Recreationally active males and females: Subjects to be considered recreationally must regularly engage in >150 min/wk of physical activity (e.g., resistance training, sport or activity specific exercise, group exercise, or aerobic exercise). Healthy participants, defined as not currently injured, or recovering from an injury within the past 12 months, or undergone surgery within the last 12 months, or with any known history of moderate to severe traumatic brain injury resulting in impaired judgment or inability to make sound decisions or mild traumatic brain injury (mTBI, also commonly named "concussion") within the last 12 months.
  Interventions: Diagnostic Test: Multimodal Assessment
- Athletes or performing artists with reported history of concussion: Participants will be considered if they are recreationally active or considered an athletic performer (i.e.,history of participation in athletics at the university, amateur, elite or professional levels, or a military veteran), or a performing artist (i.e., stunt actors, circus artists, dancers or acrobats) with reported history of concussion incident(s), with most recent incident occurring >1 month and less than five years from the study testing dates.
  Interventions: Diagnostic Test: Multimodal Assessment

INTERVENTIONS:
Diagnostic Test: Multimodal Assessment — Participants will complete BISQ/health questionnaire and proceed to each testing station with 15 minute rest breaks in between randomly ordered assigned stations.
  Other Names: Immediate Post-Concussion and Cognitive Testing (ImPACT); Sport Concussion Assessment Tool (SCAT 5); Brain Injury Screening Questionnaire (BISQ); Combined Functional near-infrared spectroscopy (fNIRS) with external kinematic sensors +modified Balance Error Scoring System (mBESS) and modified Dynamic Gait Index (mDGI) _ cognitive tasks

SUMMARY:
This study aims to explore possible solutions needed for valid and reliable multidimensional objective assessment tools to use in screening performers for concussions, as well as, for use postinjury assessment and management of the mild traumatic brain injury, regardless of time since injury occurrence. These mobile tools would also enable clinicians to test the effectiveness of the interventions used post-concussion, prior to fully releasing the performer back into full performance/active status.

DETAILED DESCRIPTION:
Participants will have study benefits and risks explained to them and after consent has been obtained each participant will be assigned an Identification number and attend their assigned testing day.

Testing day will consist of completing a seven page clinician-created medical-health questionnaire to determine that they are free of cardiovascular, metabolic, psychiatric or neurologic disease, do not have cognitive or substance-abuse problems or are taking any medications that may impair cognition, balance or functional mobility such as gait.

Participants will also complete the Brain Injury Screening Questionnaire (BISQ, Mount Sinai School of Medicine, New York, NY) to additionally screen for lifetime history of traumatic brain injury (TBI) and reduce consequences of undiagnosed mTBI.

Tests will then be conducted in three parts. First, to evaluate neuromotor and neurocognitive abilities, participants will complete a modified balance error test and a modified version of the dynamic gait index without and with additional cognitive tasks. These tests will be performed while wearing external sensors recording kinematic data and a (wearable) functional near-infrared spectroscopy cap system (NIRSport1) unit monitoring brain tissue oxygenation and perfusion.

Second test that the above multimodal test will be compared to is the sport concussion assessment tool (SCAT 5).

The third test conducted and used to compare the multimodal approach to will be the Immediate post-concussion and cognitive testing (ImPACT).

Participants will be allotted a 15-minute break period between each test.

ELIGIBILITY:
Inclusion Criteria:

* Recreationally healthy and active or considered an athletic performer, males and females, to regularly engage in >150 min/week of physical activity.
* Participants considered an athletic performer if they have history of participating in athletics at the university, amateur, elite or professional level, or are a military veteran.
* Healthy participants defined as not currently injured, or recovering from an injury within the past 12 months, or undergone surgery within the last 12 months, or with any known history of moderate to severe traumatic brain injury resulting in impaired judgement or inability to make sound decisions within the last 12 months.
* Post concussion participants are eligible if their last concussive event occurred within a month and up to 5 years of the date of data collection.

Exclusion Criteria:

* If younger than 18 or >50 years of age.
* Current cardiovascular, metabolic, psychiatric, or neurologic disease or cognitive or substance-abuse problems or taking medications that may impair cognition, balance, or functional mobility such as gait.

Ages: 18 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: 50 male and female athletes and performers will be invited to participate.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-05 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Proof of concept for the use of multimodal objective measures for mTBI assessment & treatment guide | 3-6 months for data acquisition and data analysis
  Demonstrate functional objective measures can be used regardless of time since injury to provide improved clinical diagnosis, determinant of injury, remanence of injury events still occurring

SECONDARY OUTCOMES:
Advanced portability of functional objective testing in concussion | 3-6 months for data acquisition and data analysis
  Exploration of combined wearable tools to provide functional objective data that better reflect brain activity and possible impairments post concussion throughout brains recovery

CONTACTS AND LOCATIONS:
Locations (1):
- California State University, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No